CLINICAL TRIAL: NCT01535573
Title: Clinical Trial of Serotonin Medication Combination in Cocaine Dependence
Brief Title: Citalopram for Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joy Schmitz (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Joy Schmitz, Professor , Behavioral Sciences, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2P50DA009262-16A1 (NIH); 2P50DA009262-16A1 (NIH)
Record Dates: First submitted 2011-10-24; First posted 2012-02-17 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; citalopram; treatment; serotonin
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Citalopram low dose (Active Comparator): Citalopram 20 mg
  Interventions: Drug: Citalopram
- Citalopram high dose (Active Comparator): Citalopram 40 mg
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — 20 mg once per day for 9 weeks
  Arms: Citalopram low dose
Drug: Citalopram — 40 mg per day for 9 weeks
  Arms: Citalopram high dose
Drug: Placebo — 0 mg per day for 9 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2 clinical trial of citalopram pharmacotherapy for treatment of cocaine dependence. Using a double-blind, randomized controlled design, eligible cocaine dependent patients will be assigned equally to one of three medication conditions: placebo or the Selective serotonin re-uptake inhibitor (SSRI) agent, citalopram at either 20 mg per day or 40 mg per day. It is hypothesized that citalopram will reduce cocaine use and increase periods of sustained abstinence substantially more than placebo. Performance on a set of behavioral tasks of impulsivity will be analyzed as potential predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 60 years of age
* meet Diagnostic and Statistical Manual 4 (DSM-IV) criteria for current cocaine dependence
* be in acceptable health on the basis of interview, medical history and physical exam
* able to provide the names of at least 2 persons who can generally locate their whereabouts.

Exclusion Criteria:

* diagnosis of any psychoactive substance dependence other than cocaine, marijuana, or nicotine
* have a psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
* medical conditions contraindicating citalopram pharmacotherapy
* taking medications known to have significant drug interactions with the study medication
* pregnant or nursing for female patients
* having plans to leave the immediate geographical area within 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, Ph.D., Principal Investigator — University of Texas at Houston
Locations (1):
- UT-Houston Behavioral and Biomedical Sciences Building, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
Started | 21 | 44 | 43
Completed | 13 | 23 | 24
Not Completed | 8 | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo | Total
Number analyzed (Participants) | 21 | 44 | 43 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.905 (7.578) | 44.477 (9.488) | 47.116 (8.724) | 46.000 (8.846)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 8 | 19
  Male | 18 | 36 | 35 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 0 | 1
  Black or African American | 18 | 32 | 31 | 81
  Hispanic | 2 | 5 | 5 | 12
  White | 1 | 6 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 21 | 44 | 43 | 108
Number of Years of Education [Mean (Standard Deviation); unit: years] | 12.571 (2.216) | 12.045 (1.796) | 12.488 (1.921) | 12.324 (1.932)
Number of Days of Cocaine Use in Past 30 Days [Mean (Standard Deviation); unit: days] | 12.238 (2.216) | 17.114 (9.163) | 14.465 (9.815) | 15.111 (8.594)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Cocaine Abstinent During the Last 2 Weeks of Treatment (Weeks 8-9), as Assessed by Urine Test
Description: Urine samples were tested for benzoylecgonine, which is a metabolite of cocaine that is excreted in the urine. The presence of benzoylecgonine in the urine indicates cocaine use.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
Number analyzed (Participants) | 21 | 44 | 43
Participants | 0 | 4 | 2

2. Secondary Outcome: Proportion of Cocaine-positive Urines Per Week
Description: Mean proportion of cocaine-positive urines per week, averaged across 9 weeks, is reported. Urine was collected three times each week over 9 weeks. Missing data is imputed as cocaine use.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: proportion of cocaine urines per week
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
Number analyzed (Participants) | 21 | 44 | 43
proportion of cocaine urines per week | 0.85 (0.23) | 0.8 (0.3) | 0.85 (0.25)

3. Secondary Outcome: Number of Participants With Cocaine-negative Urines Collected During Treatment Period
Description: as for outcome 1
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
Number analyzed (Participants) | 21 | 44 | 43
Participants | 14 | 26 | 27

4. Secondary Outcome: Retention as Assessed by Number of Participants Remaining in Treatment
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
Number analyzed (Participants) | 21 | 44 | 43
Participants | 13 | 23 | 24

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Citalopram Low Dose | Citalopram High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/44 | 1/43
Other Adverse Events (participants affected / at risk) | 9/21 | 20/44 | 10/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram Low Dose (N=21) | Citalopram High Dose (N=44) | Placebo (N=43)
Hospitalization for Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram Low Dose (N=21) | Citalopram High Dose (N=44) | Placebo (N=43)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal electrocardiogram (EKG) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Drowsiness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Not Sleeping Well (General disorders) | 2 (2) | 1 (4) | 4 (8)
Headache (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nervousness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blurry Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Increased Urination (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Change in Sexual Function (General disorders) | 0 (0) | 2 (3) | 0 (0)
Sweating (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Difficulty Walking (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Loss of Appetite (General disorders) | 1 (1) | 4 (6) | 0 (0)
Confusion (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes